CLINICAL TRIAL: NCT01666093
Title: NON-HEALING ULCERS WITHOUT CRITICAL LIMB ISCHEMIA (NEWLI-Trial): A Single Center Pilot Trial on the Efficacy of an Endovascular Approach for Treatment of Non-healing Lower Limb Ulcers in Patients Presenting With a Mild to Moderate Peripheral Artery Disease
Brief Title: Non-Healing Ulcers Without Critical Limb Ischemia
Acronym: NEWLI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Robert F Bonvini, MD, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEWLI-Trial; NAC 12-025 (Other: CER : 12-054)
Record Dates: First submitted 2012-08-09; First posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Peripheral Artery Disease Without Critical Limb Ischemia
Keywords: peripheral artery disease; endovascular procedure; non-healing ulcer
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- revascularization group (Other): patients will revascularized after a conservative treatment failure of at least 4 weeks
  Interventions: Procedure: Angioplasty of the lower limbs vessels

INTERVENTIONS:
Procedure: Angioplasty of the lower limbs vessels — Standard revascularization techniques will be used in the study

SUMMARY:
Background: Lower limb arterial revascularization procedures, either percutaneously or surgically performed, are an established treatment modality of ischemic foot ulcers, especially in the setting of a critical limb ischemia. Many other lower limb ulcers are secondary to a combined disease, which may include a concomitant venous disease (chronic venous insufficiency or varicous disease) or a micro-angiopathic disease (i.e. small vessel disease). In this setting, and especially in the absence of a concomitant severe macro-angiopathic disease, the safety and efficacy of a percutaneous lower limb revascularization have so far never been evaluated in a prospective study.

Aim: This study is aimed to evaluate the safety and the efficacy of an endovascular revascularization approach of the lower limb, in all consecutive patients presenting with a non-healing ulcer associated with a mild to moderate peripheral artery disease (i.e. mixed-origin ulcers).

Material and methods: This prospective study will consecutively include all patients presenting with a non-healing ulcer. Included patients must have all the concomitant ulcer co-factors being adequately treated for at least 6 months. Accordingly, an underlying venous disease, infectious disease or inflammatory disorder must be previously evaluated and adequately treated (i.e. compression stocking, varices stripping, antibiotics, local ± systemic anti-inflammatory, etc.). Furthermore, a non-invasive arterial evaluation must be obtained in all patients. The arterial screening must included an ankle-brachial index (ABI) and toe pressure (TP) measurements, a trans-cutaneous oxygen measurement (tcPO2) at the foot and calf levels and a non-invasive arterial mapping (i.e. angio-CT or angio-MRI). This arterial work-up must be compatible with the presence of a mild to moderate peripheral artery disease without any sign or criteria suggesting the presence of a critical limb ischemia.

End-points: The success rate of perform an endovascular revascularization intervention in all consecutive patients which qualify according to the inclusion criteria (technical feasibility). Establish the proportion of procedural related complications (safety). Analyze the clinical and the para-clinical improvements in term of heal of the ulcers, as well as the improvement of the ABI, TP, tcPO2 at 1 week, 1-3-6 months after the procedure (efficacy).

Sample size: The investigators plan to include ≈ 30 patients in two years. After 1 year of enrollment the investigators will perform an interim analysis and will decide at that moment, according to the observed end-points, if prolonging the study would be of any scientific value or if the study has to be interrupt earlier because of a significant improvement of all already treated ulcers.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

1. Patients need to be at least 18 years old
2. Patients have to be admitted to the university hospitals of Geneva for a non-healing lower limb ulcer.

   - Eligible patients are those presenting with non-healing lower limb ulcers for more than 3 months.
   * Patients will be hospitalized in the Dermatology inpatient clinic.
   * Patients had to benefit from at least one thin skin autograft at the ulcer level in the past or during the index hospitalization.
3. Before inclusion in the study, patients must undergo complete angiological diagnostic work-up including:

   * A baseline ABI, toe pressure and tcPO2 measurements,
   * A non-invasive arterial imaging including an angio-CT scan or an angio-MRI,
4. The non-invasive arterial work-up must revel mild to moderate PAD, without any criteria or sign of CLI (see flow-chart):

   * Ankle pressure ≥ 50 mmHg,
   * + ABI: < 0.9 or > 1.3,
   * ± Toe pressure : 30-100 mmHg
   * ± tcPO2: 20-40 mmHg,
   * At this moment the patient may be included in the study protocol.
5. All patients presenting with mild to moderate PAD and evidence of at least 1 impaired arterial vessel targeting the ulcer will initially undergo conservative impatient clinic care for at least 2-4 weeks and benefit from at least 1 thin skin autograft.

   * Persisting surface of lower limb ulcers will be assessed 1 month later:

     -- In the presence of a healed ulcer surface > 70%, the patient will undergo 6 months of clinical follow up at 1-3-6 months.

     1. In case of persistence of healed ulcer surface > 70% clinical success will be achieved.

     2. In presence of healed ulcer surface < 70% the patient will undergo a new angiological work-up.
   * If mild to moderate PAD will be again outlined the patient will join the < 70% healed ulcer group.
   * On the other hand, if CLI will be pointed out lower limb revascularisation and at least one thin skin autograft will be performed.

     -- In presence of a healed ulcer surface < 70%, endovascular PTA and at least one thin skin autograft will be performed. The ulcers healing will then be monitored at 1-3-6 months and persisting ulcers surface re-assessed:
   * in presence of an healed ulcer surface > 70% clinical success will be achieved,
   * if presence of an healed ulcer surface < 70% clinical failure will be retained.

Exclusion Criteria:

1. Patients who refused to give their written informed consent.
2. Patients, in whom the angiological work-up shows the presence of a CLI, mandating a revascularization procedure attempt (i.e. ankle pressure < 50mmHg, toe pressure < 30mmHg, tcPO2 < 20mmHg) (see particular situation n°2).
3. Patients who do not present with peripheral artery disease (i.e., ABI > 0.9 - < 1.3, TP > 100mmHg, tcPO2 > 40mmHg).
4. Patients in whom the angiological-dermatological work-up shows the presence of another reversible cause of the non-healing ulcer:

   - Special attention will be given to the presence of a treatable venous insufficiency (e.g. compression stocking, varices stripping), an underlying inflammatory/infectious process (treatable with antibiotics or topic-systemic antiinflammatory medications) or other reversible mechanical factors (unadapted shoes, etc.).
5. Patients without any significant lesion of the arterial tree (ilio-femoro-popliteal and infra-popliteal):

   - In case there will be a single BTK vessel disease not perfusing the ulcer area (e.g. pre-tibial ulcer with a significant stenosis of the posterior tibial artery which does not perfuse the ulcer region), the patient will not be included in the study because any significant ulcer improvement would be expected from this non-target vessel revascularization.
6. Patients in whom the scheduled revascularization procedure will be judged too risky for the patient's safety:

   * Chronic kidney failure (= Creatinin Clearance < 20ml/min) with an increased risk of contrast induced nephropathy,
   * Too complex arterial disease or anatomy, in which the estimated procedural technical success rate is < 50% (i.e. complex chronic total occlusion).
7. Patients in whom an amputation is unavoidable, despite any revascularization attempt (e.g. extensive skin necrosis [Rutherford class 6]), - If, it will be estimated that, a successful revascularization procedure may reduce the level of amputation, or if a successful intervention may improve the amputation's healing process, the patient may be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Ulcer healing | at 6 months
  1) Procedural efficacy: efficacy will be evaluated according to clinical and para-clinical parameters:
  a. Clinical efficacy: i. ulcer heal or improvement at 6 months; ii. avoidance of minor (i.e. toe or for-foot) or major (i.e. below or above the knee) amputations; iii. improvement of the ulcer-related pain:
  1. The ulcer-related pain will be evaluated with the use of the Borg visual assist scale (Borg VAS) before, at 1 week, 1-3-6 months after the procedure.
  iv. Improvement of the ulcer size:
  1. The ulcer size will be recorded by measurements and photographic records before, at 1 week, 1-3-6 months after the procedure.
  v. The number of skin grafts necessary to heal the ulcer will be recorded and compared to the number of the skin grafts which have failed to heal the ulcer in the pre-revascularization period.

SECONDARY OUTCOMES:
Efficacy | 6 months
  1. Para-clinical efficacy: improvement of the ABI, TP, tcPO2 values at 1 week, 1-3-6 months after the procedure.
  2. Procedural success, defined as a successful endovascular revascularization procedure, in all consecutive patients according to the inclusion and exclusion criteria = technical feasibility.
Safety | 6 months
  3) Procedural safety, defined as the proportion of procedures performed in the absence of any procedural-related complications (= safety).

CONTACTS AND LOCATIONS:
Locations (1):
- Angiology and Dermatology Divisions / HUG, Geneva, Canton of Geneva, Switzerland